CLINICAL TRIAL: NCT05464784
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Efficacy of MN-001 in Patients Diagnosed With Non-alcoholic Fatty Liver Disease, Type 2 Diabetes Mellitus, and Hypertriglyceridemia
Brief Title: MN-001 in Non-alcoholic Fatty Liver Disease, Type 2 Diabetes Mellitus, and Hypertriglyceridemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MN-001-NATG-202
Record Dates: First submitted 2022-06-28; First posted 2022-07-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus, Type 2; Hypertriglyceridemia; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertriglyceridemia; Non-alcoholic Fatty Liver Disease | interventions — 4-(6-acetyl-3-(3-(4-acetyl-3-hydroxy-2-propylphenylthio)propoxy)-2-propylphenoxy)butyric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MN-001 (Experimental)
  Interventions: Drug: MN-001
- MN-001 Placebo (Placebo Comparator): The placebo comparator is a tablet identical in appearance to MN-001.
  Interventions: Drug: MN-001 placebo

INTERVENTIONS:
Drug: MN-001 — MN-001 is a novel, orally bioavailable small molecule compound
  Arms: MN-001
Drug: MN-001 placebo — The placebo tablet is identical in appearance to the MN-001 tablet, and contains excipients of MN-001.
  Arms: MN-001 Placebo

SUMMARY:
The design of the Phase 2 clinical trial includes the following elements:

* Multi-center, two-arm, randomized, double-blind, placebo-controlled trial to evaluate MN-001 (tipelukast) vs. placebo in approximately 40 patients in the U.S.
* Patients will be randomized 1:1 to receive either 500 mg/day of MN-001 (tipelukast) or placebo for 24 weeks.
* The co-primary endpoints are (1) change from baseline in liver fat content measured by controlled attenuation parameter (CAP) score at Week 24, and (2) change from baseline in fasting serum triglycerides at Week 24. FibroScan® is a non-invasive, quantitative, and accurate measure of liver fat content commonly used in early phase trials to measure treatment response.
* Secondary endpoints include safety and tolerability and changes in lipid profile (HDL-C, LDL-C, and total cholesterol).

ELIGIBILITY:
Inclusion Criteria:

* FibroScan® CAP score ≥ 248 dB/m within 8 weeks of randomization.
* Diagnosis or history of Type 2 Diabetes mellitus with hemoglobin A1c (HbA1c) >6.5 and ≤10% at Screening.
* Fasting serum triglycerides (TG) at Screening >150 mg/dL
* On a stable dose of oral antidiabetic therapy for a minimum of 3 months prior to Screening.

Exclusion Criteria:

* Other causes of chronic liver disease (autoimmune, primary biliary cholangitis, HBV, HCV, Wilson's, α-1-antitrypsin deficiency, hemochromatosis, biopsy-proven cirrhosis, hepatocellular carcinoma);
* Documented history of advanced liver fibrosis
* Evidence of cirrhosis, hepatic decompensation, portal hypertension including splenomegaly, ascites, encephalopathy and/or esophageal varices;
* Diagnosis or history of Diabetes mellitus type 1;
* Weight change >5% within last 3 months of Screening visit;
* Active gastrointestinal disease or history of gastric bypass surgery which could interfere with the absorption of oral medication;
* History of clinically significant acute cardiac event within 6 months of Screening;

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in controlled attenuation parameter (CAP) score by sound-based elastography at Week 24 | Week 24
Mean change from baseline in fasting serum triglyceride levels at Week 24 | Week 24

SECONDARY OUTCOMES:
Safety and tolerability of MN-001 | Baseline to Week 24
  Incidence of adverse events, abnormal clinical laboratory results
Mean change from baseline in lipids | Baseline to Week 24
  Changes in lipids (HDL-C, LDL-C, total cholesterol) after MN-001 treatment for 24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Jubilee Clinical Research, Inc., Las Vegas, Nevada
  - Pinnacle Clinical Research at South Texas Research Institute, Edinburg, Texas

IPD SHARING:
Plan to Share IPD: No